CLINICAL TRIAL: NCT05949554
Title: Characterization of Electroencephalographic (EEG) Signatures of Chronic Pain Patients Receiving Intravenous Ketamine.
Brief Title: Electroencephalographic (EEG) Profils for Patients on Intravenous Ketamine.
Acronym: KetEEG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); M3DISIM (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230352; 2023-A00080-45 (Other: IDRCB)
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Neuropathic Pain
Keywords: Pain medicine; EEG biomarkers; Refractory neuropathic pain; Ketamine
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ketamine infusion — Continuous measurement of burst suppression (BS) (%) and 95% spectral frequency front (SEF95) on frontal EEG Sedline® Masimo Corporation, USA).
  EEG recording will start 10 minutes before the beginning of infusion until the total amount of 10 milligrams of Ketamine has been infused.
  The duration varies depending on patient's weight.
  Each patient will receive a dose of 0,5 mg/kg over a period of time of 2 or 4 hours.

SUMMARY:
Chronic pain symptoms can lead to sleep and mood disorders, restrict domestic and work activities and have a significant impact on quality of life. The prevalence of chronic pain in the general population varies between 10 and 52% depending on the study, 7% of which is neuropathic pain.

Anxiety-depression comorbidities are found in a large number of patients, with harmful consequences on pain since they exacerbate symptoms and their repercussions. Conversely, pain increases psychological distress.

Ketamine has been used in the context of depressive episodes for its rapid action. It is also increasingly used in chronic pain due to its ability to regulate the "wind-up" effect, a phenomenon involved in the central hypersensitization that is inevitably present in neuropathic pain of prolonged duration.

Several studies have found electroencephalographic (EEG) signatures associated with a good antidepressant response to Ketamine. The frequency, absolute and relative power and cordance of the EEG signal in certain frequency ranges (theta, alpha, beta and gamma) could be useful to guide and adapt therapies for depression and pain.

DETAILED DESCRIPTION:
The prevalence of chronic pain in the general population varies between 10 and 52% depending on the study, 7% of which is neuropathic pain. These neuropathic pains have various origins: post-surgical, post-herpetic, post-traumatic, etc. These chronic pain symptoms can lead to sleep and mood disorders, restrict domestic and work activities and have a significant impact on quality of life.

Anxiety-depression comorbidities are found in a large number of patients, with harmful consequences on pain since they aggravate symptoms and their repercussions. Conversely, pain increases psychological distress.

Ketamine, derived from phencyclidine, is an anesthetic agent used since the 1960s. It acts by non-competitive antagonism of the N-methyl-D-aspartate (NMDA) receptors found mainly in the hippocampus and prefrontal cortex. This receptor is one of the binding sites for glutamate, an excitatory neurotransmitter involved in the transmission of painful messages, long-term memory processes, and hyperalgesia. Ketamine has been used in the context of depressive episodes characterized by its rapid action. It is also increasingly used in chronic pain due to its regulating action on the "wind up" effect, a phenomenon involved in the central hypersensitization that is inevitably present in neuropathic pain with a prolonged course. The mechanisms underlying the improvement of neuropathic pain after ketamine infusion are not fully elucidated. Some animal studies suggest a prolonged anti-aversive effect on the anterior cingulate cortex or a weaker connectivity between the prefrontal cortex and the precuneus in patients who respond to ketamine. At the same time, the antidepressant effect seems to be linked to an action on the prefrontal cortex. Overall, the literature shows a strong association between anxiety-depressive symptoms and chronic pain.

EEG recording of patients with neuropathic pain before and during ketamine infusion would allow the acquisition of important electro-physiological data.

Several studies have found that EEG signatures was associated with a good antidepressant response to Ketamine. The frequency, absolute and relative power and cordance of the EEG signal in certain frequency ranges (theta, alpha, beta and gamma) could be useful for guiding and adapting therapies for depression as well as pain.

Patients over 18 years old are eligible to participate in this protocol. At the time of the pain follow-up consultation, they will be given a letter of information on the objectives and progress of the study. Their non-opposition to participate in this study will be collected at the time of their entry into the department as part of their scheduled hospitalization.

The protocol will start during a scheduled hospitalization to administer the first Ketamine infusion.

The protocol does not interact with the care procedure.

- During their hospitalization, the participants would have to complete of a concise pain questionnaire and Hospital Anxiety and Depression scale (HAD score).

Before Ketamine infusions at week 1 (W1) and week 3 (W3), concise pain questionnaire, HAD score, Pain Catastrophizing Scale (PCS score), and the Montreal Cognitive assessment (MoCA test) are performed. Then, an EEG is recorded for about 60 minutes using a noninvasive device (Masimo ©).

The study physician collecting the data was not involved in the patient's management at any time. The measures cannot influence the prescribing physician since at this stage the data are not yet analyzed and available.

No added risk.

Continuous data will be expressed as median [interquartile] and categorical data as n (%). Categorical variables will be compared by Mann-Whitney test and continuous variables by Wilcoxon test.

The correlation between pain, anxiety-depressive symptoms and catastrophizing will be estimated by Pearson correlation test.

The ability of the various EEG parameters of interest to predict the occurrence of an improvement in pain will be estimated by constructing a ROC curve. The area of these ROC curves will be measured, and the corresponding 95% confidence interval estimated. The areas under the ROC curve of the different parameters will be compared by DeLong test.

The statistical analysis will be carried out using the statistical analysis software " R " (The R Foundation, Vienna, Austria) under the responsibility of Pr Etienne GAYAT.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Eligible for Ketamine infusions in the context of chronic pain refractory to usual therapies
* Patient informed and having expressed his non-objection to participation in this research
* Patient who is not subject to a legal protection measure

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with a contraindication to ketamine.
* Patient opposed to protocol participation
* Pregnant woman
* Patient under legal protection
* Patient not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 or over hospitalized for Ketamine infusion in the context of neuropathic pain in the Department of Pain Medicine at Lariboisière Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Characterizing the EEG signature of chronic pain patients before and during intravenous Ketamine infusion | Week 3
  Analysis of EEG changes by calculating absolute and relative power and cordance of the EEG signal in certain frequency ranges at different times of the infusion before and during Ketamine infusion at W1 and W3 EEG recording and its changes before and during Ketamine infusion at W1 and W3.

SECONDARY OUTCOMES:
To establish a correlation between improvement in pain after ketamine and anxiety-depressive symptoms. | Week 3
  For all patients, anxio-depressive symptoms assessed by the Hospitality Anxiety and Depression (HAD) scale.
To characterize the EEG signature of chronic pain patients in different subgroups as depressed and catastrophism | Week 3
  Catastrophism related pain assessed by Pain Catastrophism Scale (PCS)
To establish the absence of cognitive dysfunction after infusion of Ketamine. | Week 3
  Psychometric testing with the MoCA (Montreal Cognitive Assessment) psychometric scale and the MemScreen
To characterize the EEG signature of chronic pain patients in different subgroups as depressed and catastrophism | Week 3
  Pain assessment by the concise pain questionnaire validated in French. A score above 7 points attests to the presence of anxiety-depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice VALLEE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris, Lariboisière Hospital, Department of Anesthesiology and Intensive Care; Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris, Lariboisière Hospital, Department of Anesthesiology and Intensive Care